CLINICAL TRIAL: NCT00367484
Title: Multicentre, Single Arm, Open, Phase IV Study To Evaluate Immunogenicity And Safety Of Subcutaneous r-hIFN Beta-1a (Rebif®) Using Clone 484-39 In The Treatment Of Relapsing Remitting Multiple Sclerosis
Brief Title: Study To Evaluate The Immunogenicity And Safety Of r-hIFN Beta-1a (Rebif®) Using Clone 484-39 In Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24810
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Results first posted 2010-08-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

ARMS (1):
- Rebif® (clone 484-39) (Experimental): Rebif® 44 mcg, three times per week (tiw), subcutaneously (s.c.) During the first 4 weeks of the study, subjects underwent a dose titration regimen of 40% of Rebif® 22 mcg or 20% of Rebif® 44 mcg tiw (8.8 mcg per injection) in the first and second week followed by 100% of Rebif® 22 mcg or 50% of Rebif® 44 mcg (22 mcg per injection) in the third and fourth week. After 4 weeks, subjects received 44 mcg injected s.c. tiw.
  Interventions: Biological: Rebif® (clone 484-39)

INTERVENTIONS:
Biological: Rebif® (clone 484-39) — s.c. administered Rebif®
  Other Names: Recombinant-human interferon beta-1a; r-hIFN Beta-1a

SUMMARY:
The objectives of the study are:

- comparison of the incidence and time course of the development of neutralizing antibodies (NAbs) to Rebif after 48 weeks of therapy, to historical data from Serono clinical trial databases to assess the safety and tolerability of Rebif®

ELIGIBILITY:
Inclusion Criteria:

* Have multiple sclerosis (MS) with two or more relapses in the past two years and is eligible for interferon therapy.
* Be between 18 and 60 years of age, inclusive.
* Have given written informed consent, prior to any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.
* Be willing and able to follow all study procedures for the duration of the study.
* Have an Expanded Disability Scale Score (EDSS) less than 6.0
* If female, she must either

  1. be post menopausal or surgically sterilised; or
  2. use a hormonal contraceptive, intra uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and
  3. be neither pregnant nor breast feeding. Confirmation that the subject is not pregnant must be established by a negative SERUM human Chorionic Gonadotrophin (hCG) pregnancy test between 28 to 7 days before Study Day 0.Urine pregnancy test must be done if serum hCG pregnancy test was performed more than 7 days before Study Day 0. A pregnancy test is not required if the subject is post menopausal or surgically sterilised.

Exclusion Criteria:

* Prior Interferon beta therapy (either beta-1b or beta-1a).
* Major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol.
* Significant immunosuppressive therapy within the 6 months prior to enrolment.
* Known history of hypersensitivity to natural or recombinant interferon beta, human serum albumin, or any other component of the formulation.
* Epilepsy with a history of seizures not adequately controlled by treatment.
* Have greater than Grade 1 toxicity for liver function tests (Aspartate Transaminase (AST), Alanine Transaminase (ALT), Gamma-Glutamyl Transferase (GGT) or total bilirubin) at the Screening visit
* Have significant leukopenia (greater than Grade 1 toxicity for total white blood cell count or lymphopenia) at the Screening visit
* Have had treatment with oral or systemic corticosteroids or Adrenocorticotrophic hormone (ACTH) within 1 month of the Screening visit or between the screening visit and study day 0.
* Cytokine or anti-cytokine therapy within the 3 months prior to the Screening visit or between the screening visit and study day 0.
* Use of immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporin, methotrexate, azathioprine, linomide) within the 6 months prior to the Screening visit or between the screening visit and study day 0.
* Have taken intravenous immunoglobulin or glatiramer acetate or mitoxantrone or any investigational drug or experimental procedure within the 3 months prior to the Screening visit or between the screening visit and study day 0.
* Prior use of cladribine or have received total lymphoid irradiation.
* Presence of systemic disease that might interfere with patient safety, compliance or evaluation of the condition under study (e.g. poorly controlled insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, human immunodeficiency virus (HIV), human T-lymphotrophic virus 1 (HTLV-1)).

Other concurrent systemic disorders incompatible with the study (at the Investigator's discretion).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Stubinski, M.D., Study Director — Merck Serono SA - Geneva

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened for enrollment from 27 May 2004 and attended the last visit on 30 January 2006. Four hundred and eighty four subjects were screened for enrollment and 460 were enrolled. Two subjects (0.4%) were excluded from the ITT Population since they had no post-Baseline NAb assessment due to withdrawing from the study prematurely.
Pre-assignment Details: At Week -4 (to Week -1), subjects provided written informed consent and underwent screening procedures. Twenty four subjects were not included in the study: the reasons were "Not met all eligibility criteria" (18 subjects) and "Other" (6 subjects)
Groups:
- Rebif® (Clone 484-39): subcutaneously administered Rebif® 44mcg three times per week
Period: Overall Study
Arm/Group | Rebif® (Clone 484-39)
Started | 460
Completed | 443 (Safety population = 460 Intent To Treat (ITT) population = 458)
Not Completed | 17
Not completed — Adverse Event | 7
Not completed — Withdrew informed consent | 5
Not completed — Travel to USA | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — The choice of the patient | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rebif® (Clone 484-39)
Number analyzed (Participants) | 458
Age, Categorical [Count of Participants; unit: Participants] — ITT population
  Participants
    <=18 years | 0
    Between 18 and 65 years | 458
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — ITT population
  years | 36.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population
  Participants
    Female | 336
    Male | 122
Region of Enrollment [Number; unit: participants] — ITT population
  participants
    Estonia | 36
    France | 2
    United Kingdom | 13
    Hungary | 23
    Lithuania | 69
    Morocco | 5
    Poland | 69
    Romania | 87
    Russian Federation | 43
    Serbia | 80
    Tunisia | 31
Neutralising Antibody (NAb) Status [Number; unit: Participants not testing NAb positive] — Participants who did not test positive for NAb at baseline. The NAb+ value was defined as NAb ≥ 20 NU/ml.
  Participants not testing NAb positive | 458

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Testing Positive for Neutralising Antibody (NAb)
Description: Participants who were NAb+ at 48 weeks (or at the last available NAb assessment up to Week 48). The NAb+ value was defined as NAb ≥ 20 NU/ml.
Time Frame: 48 Weeks
Population: Intent To Treat (ITT) population, Last Observation Carried Forward (LOCF)
Measure: Number; unit: NAb+ participants
Arm/Group | Rebif® (Clone 484-39)
Number analyzed (Participants) | 458
NAb+ participants | 73

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Comprehensive assessments of any apparent toxicity experienced by the subject were performed throughout the course of the study. Study site personnel reported any AE, whether observed by the Investigator or reported by the subject.
Arm/Group | Rebif® (Clone 484-39)
Serious Adverse Events (participants affected / at risk) | 11/460
Other Adverse Events (participants affected / at risk) | 378/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif® (Clone 484-39) (N=460)
Pneumonia (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Injection site abscess (Infections and infestations) | 1 (1)
Injection site cellulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif® (Clone 484-39) (N=460)
Influenza like illness (General disorders) | 188 (284)
Injection site erythema (General disorders) | 67 (71)
Pyrexia (General disorders) | 50 (57)
Fatigue (General disorders) | 37 (40)
Chills (General disorders) | 35 (39)
Asthenia (General disorders) | 29 (35)
Headache (Nervous system disorders) | 129 (208)
Upper respiratory tract infection (Infections and infestations) | 37 (45)
Influenza (Infections and infestations) | 32 (58)
Urinary tract infection (Infections and infestations) | 27 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 43 (53)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (36)
Nausea (Gastrointestinal disorders) | 24 (26)
Alanine aminotransferase increased (Investigations) | 25 (26)
Insomnia (Psychiatric disorders) | 31 (34)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 40 (53)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 36 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other